CLINICAL TRIAL: NCT03611816
Title: Biological Bank for Studies Related to Atrial Fibrillation and Stroke
Brief Title: Biological Bank for Atrial Fibrillation and Stroke
Acronym: BAFA
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0538; 2017-A03327-46 (Other: ID-RCB)
Record Dates: First submitted 2018-01-31; First posted 2018-08-02 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1a: Patient with atrial fibrillation and without stroke history.
  Interventions: Biological: Blood taken; Genetic: Blood taken
- Group 1b: Patient with atrial fibrillation with scheduled electrophysiology exploration or ablation.
  Interventions: Biological: Blood taken; Genetic: Blood taken
- Group 1c: Patient with atrial fibrillation and with stroke history.
  Interventions: Biological: Blood taken; Genetic: Blood taken
- Group 2: Patients aged over 80 years old and without history of atrial fibrillation.
  Interventions: Biological: Blood taken; Genetic: Blood taken
- Group 3: Patient with cryptogenic stroke or transient ischemic attack history before the age of 50.
  Interventions: Biological: Blood taken; Genetic: Blood taken

INTERVENTIONS:
Biological: Blood taken — Collection of clinical data
Genetic: Blood taken — Collection of DNA
Genetic: Blood taken — Collection of plasma
  Groups: Group 1b

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia encountered in clinical practice. This arrhythmia is responsible for 15% of strokes and more than 30% of strokes on people over 65 years.

According to studies, 30 to 40% of isolated atrial fibrillations could be familial. Atrial fibrillation has significant genetic heterogeneity. About 40 genes have been identified as potentially involved. Studies have identified genes common to the risk of atrial fibrillation and stroke. Despite the pathophysiology of atrial fibrillation has been intensively and extensively studied for almost a century, there are still many questions. The pathophysiology is not sufficiently understood to allow finding more effective therapies. It is necessary to identify genetic determinants and thus potentially new pharmacological targets more adapted.

The establishment of a biological database will test hypotheses concerning the genetic origin and thromboembolic process of atrial fibrillation and associated stroke.

ELIGIBILITY:
Group 1a

* Inclusion Criteria :

  - AF history
* Exclusion Criteria :

  * No AF history
  * patient who didn't signed consent

Group 1b

* Inclusion Criteria :

  * AF history
  * Scheduled electrophysiological exploration or AF ablation
* Exclusion Criteria :

  * No AF history
  * pregnant women
  * patient who didn't signed consent

Group 1c

* Inclusion Criteria :

  * AF/AT history
  * Stroke history
* Exclusion Criteria :

  * No Stroke history
  * patient who didn't signed consent

Group 2

* Inclusion Criteria :

  * patient over 80
  * ECG: sinusal rhythm
  * TTE : no left atrial dilatation
* Exclusion Criteria :

  * atrial fibrillation history
  * TTE : Left atria >25cm², > 34m/m2), FEVG < 50%
  * ECG : QRS > 90 ms
  * cardiac pathologies (excepted hypertension and valvulopathies)
  * History of stroke and transient ischemic attack
  * patient who didn't signed consent

Group 3

* Inclusion Criteria :

  * cryptogenic stroke or transient ischemic attack history before 50 yo
  * No AF history
* Exclusion Criteria :

  * AF history
  * stroke or transient ischemic attack over 50 yo
  * patient who didn't signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial fibrillation patient Stroke patient Patient over 80
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2029-04-23 (Estimated); Study Completion 2029-04-23 (Estimated)

PRIMARY OUTCOMES:
Quality of DNA sample | 1 day (the day of the storage)
  Quality is based on the measure of the purity of DNA with absorbance assay at 260/280nm on a spectrophotometer. For Plasma sample, purity is based on absence of hemolyzed blood by visual observation.
Quality of Plasma sample | 1 day (the day of the storage)
  Quality is based on the purity of Plasma sample that is based on absence of hemolyzed blood by visual observation.
Quality of preservation of the sample | 7 years (during all the duration of the collection)
  The quality of preservation of the sample throughout the conservation duration is based on the number of freezing/thawing of each cryotube that will be notified. As weel as any interruption in the freezing process (power failure, freezer failure).

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Service neurologie Centre hospitalier Fleyriat, Bourg-en-Bresse
  - Service d'urgences Neurovasculaires - service de neurologie vasculaire , Hôpital Pierre Wertheimer, Bron
  - Service de rythmologie, hôpital cardiologique Louis Pradel, Bron
  - Service de médecine gériatrique Centre hospitalier Lyon Sud, Groupement hospitalier Sud, Pierre-Bénite
  - Hôpital des charpennes, Villeurbanne

IPD SHARING:
Plan to Share IPD: No